CLINICAL TRIAL: NCT03250520
Title: Pilot Study of the Application of Palliative Treatment in Children With Brain Stem Glioma and Recurrent High-grade Tumors in the Central Nervous System With the Nanomaterial Platinum Acetylacetonate (1% wt) Supported by Sol-gel Technology Functionalized Titania (NPt-Ca)
Brief Title: Application of Palliative Treatment in Children With Brain Stem Glioma and Recurrent High-grade Tumors in the Central Nervous System With the Nanomaterial NPt-Ca
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: Principal Investigator, Daniel Eduardo Alvarez Amado, Researcher in the Neurology Department, Hospital Infantil de Mexico Federico Gomez
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HIM 2017-072
Record Dates: First submitted 2017-06-10; First posted 2017-08-15 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Brain Tumor, Pediatric, Brainstem Glioma; Brain Tumor, Pediatric, Recurrent
MeSH Terms: conditions — Brain Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- glioma brain stem (Experimental)
  Interventions: Drug: Platinum acetylacetonate (1% wt) supported by sol-gel technology functionalized titania
- high grade recurrent brain tumor in the central nervous system (Experimental)
  Interventions: Drug: Platinum acetylacetonate (1% wt) supported by sol-gel technology functionalized titania

INTERVENTIONS:
Drug: Platinum acetylacetonate (1% wt) supported by sol-gel technology functionalized titania — Sol-gel process Pt(acac)2- F-TiO2 nanostructured material with antitumoral activity used as an alternative in the treatment of cancer tumors. The biocatalysts were prepared by the sol-gel route using the complex Pt(acac)2.
  Other Names: Pt(acac)2/Titanium dioxide (Ti02); Pt(acac)2/F-TiO2; NPt; NPt-Ca

SUMMARY:
This Protocol is a pilot, clinical interventional study to selected patients between five and fourteen years of both sexes, carriers of the diagnosis of glioma brain stem and high grade recurrent in the central nervous system tumors, in whom there has been no response to conventional-based surgery/radiation/chemotherapy treatment or whose location does not allow treatment with conventional measures, and that already have an indication for a neurosurgical palliative procedure. It will be a close pharmacovigilance on possible adverse effects related to the nanomaterial based on the profile of cisplatin (chemotherapeutic platinum derivative), since documented toxicity data are not counted for NPt-Ca. Quality of life will be documented with PedsQL Cancer Module© and tumor size by magnetic resonance brain images.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological diagnosis or MRI of the brain stem or tumor of recurrent high-grade glioma.
* Indication of palliative surgical treatment by neurosurgery.
* Good general condition, enabling the realization of surgical treatment.
* Scale Lansky > 20)
* conventional treatment (surgery, radiotherapy, and chemotherapy) failed or not applicable to the patient.

Exclusion Criteria:

* Patients with emerging infectious diseases or fever in the last 72 hours prior to placement of the NPt-Ca.
* Patients whose parents/carers do not authorize expressly the realization of procedure with knowledge of its experimental nature, are not agreed or established their commitment to meet follow-up parameters established by this Protocol.
* Patients with surgical complications prior to placement of the NPt-Ca.
* Patients in which the size and location of the lesion do not allow their surgical approach or an increase in volume by infiltration of the lesion with 3 ml of volume of NPt-Ca.
* Patient whose neurological condition do not allow the implementation of MRI without anesthesia.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Change in the quality of life using the PedsQL Cancer Module© | Preoperative and at 1.3, 6, 12, 18 and 24 months.
  Measures of the change of quality of life pre and after the administration of NPt-Ca using the questionnaire PedsQL Cancer Module©
Change in tumor size | Immediate, 1, 2, 3, 6, 8, 10, 12, 18 and 24 months.
  Change in tumor size after the administration of NPt-Ca using volumetric measures on the brain magnetic resonance.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Infantil de Mexico Federico Gomez, DF, Mexico

IPD SHARING:
Plan to Share IPD: Undecided